CLINICAL TRIAL: NCT04201561
Title: Safety and Efficacy of High Dose Inorganic seLenium for Preventing Chemotherapy Induced pEripheral Neuropathy in platINUM Sensitive Recurrent Ovarian, Fallopian, Primary Peritoneal Cancer: Phase III Randomised Controlled Trial
Brief Title: High Dose Inorganic Selenium for Preventing Chemotherapy Induced Peripheral Neuropathy
Acronym: SELENIUM
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Principal Investigator, Hee Seung Kim, Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SELENIUM trial
Record Dates: First submitted 2019-12-08; First posted 2019-12-17 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy; Recurrent Ovarian Carcinoma; Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Carcinoma
Keywords: peripheral neuropathy; recurrent ovarian cancer; high-dose inorganic selenium; sodium selenite
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Peripheral Nervous System Diseases | interventions — Sodium Selenite; Saline Solution; Sodium Chloride; Drug Therapy; Paclitaxel; Carboplatin; Bevacizumab

STUDY DESIGN:
Intervention Model Description: Patients enrolled in this study will be randomized into two groups. Patients in the control group will receive paclitaxel chemotherapy every 3 weeks for a total of 6 cycles and a dose of normal saline 40 ml every cycle before chemotherapy begins. Patients in the experimental group will receive a dose of selenium 2000 μg/40 ml instead every cycle before chemotherapy.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The patient will receive an intravenous selenium 2000 μg/40 ml dose just before chemotherapy begins every cycle (every 3 weeks for 6 cycles). Afterward, the same dose will be continued during the maintenance period if it is medically required or if the patient desires to do so.
  Interventions: Drug: sodium selenite pentahydrate; Drug: Chemotherapy
- Placebo group (Placebo Comparator): The patient will receive an intravenous normal saline 40 ml dose just before chemotherapy begins every cycle (every 3 weeks for 6 cycles). Afterward, the same dose will be continued during the maintenance period if it is medically required or if the patient desires to do so.
  Interventions: Drug: Normal saline; Drug: Chemotherapy

INTERVENTIONS:
Drug: sodium selenite pentahydrate — High-dose inorganic selenium (2000 μg/40 ml) will be administered before chemotherapy in patients assigned to the experimental group.
  Other Names: Selentab inj. A12CE02
  Arms: Experimental group
Drug: Normal saline — Normal saline (40 ml) will be administered before chemotherapy in patients assigned to the control group.
  Other Names: sodium chloride 0.9%
  Arms: Placebo group
Drug: Chemotherapy — Paclitaxel (175mg/m2), carboplatin (AUC 5.0 or 6.0) IV, and bevacizumab IV (15mg/kg) D1, every three weeks.
  Other Names: Paclitaxel, carboplatin and bevacizumab

SUMMARY:
This study aims to evaluate the safety and efficacy of high dose inorganic selenium in preventing and relieving chemotherapy-induced peripheral neuropathy (CIPN) in platinum-sensitive recurrent ovarian, fallopian, or primary peritoneal cancer patients. This study will be conducted as a phase III randomized controlled trial in platinum-sensitive recurrent ovarian, fallopian, or primary peritoneal cancer patients who are expected to undergo paclitaxel-carboplatin chemotherapy. A total of 68 patients need to be enrolled in this study. The primary objective of this study is to evaluate the frequency of chemotherapy-induced peripheral neuropathy. The secondary objectives are the evaluation of the severity of peripheral neuropathy and the quality of life to show that selenium is effective in preventing and relieving peripheral neuropathy induced by paclitaxel. Positive results in this study will lead to further studies investigating the effect of selenium on other chemotherapies that can induce peripheral neuropathy.

DETAILED DESCRIPTION:
High-dose selenium is known to reduce systemic inflammatory responses through antioxidant and anti-inflammatory effects. Selenium has also been shown in pre-clinical studies to inhibit chemotherapy-induced peripheral neuropathy through reactive oxygen species mechanisms in cells. Therefore, the investigators aimed to confirm the effect of preventing high dose intravenous selenium prior to chemotherapy and to prevent neuropathy caused by chemotherapy. In this study, the investigators will identify the frequency and severity of CIPN according to World Health Organization (WHO) criteria. Also, the investigators will assess the patient's quality of life (QoL), evaluate the effects of the administration of inorganic selenium on CIPN and QoL, and confirm the safety of high-dose selenium. I would like to.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent
2. Age: 19-80 years old
3. Complete or partial response according to Response Evaluation Criteria In Solid Tumors (RECIST) or Gynecologic Cancer Intergroup criteria in epithelial ovarian cancer, fallopian cancer, or primary peritoneal cancer patients who underwent either surgery or chemotherapy and those who have recurred cancer at least six months after chemotherapy.
4. Patients who have received paclitaxel chemotherapy for a minimum of 6 cycles and a maximum of 9 cycles
5. Eastern Cooperative Oncology Group performance status 0-2
6. Patients with no other concurrent disease affecting overall survival
7. Patients with normal hematologic, renal, and liver functions
8. Patients who understand the contents of the clinical trial and are capable of participating until the end of the trial

Exclusion Criteria:

1. Pregnancy or breastfeeding
2. Patients diagnosed with recurrent ovarian cancer, fallopian cancer, or primary peritoneal cancer who received secondary debulking surgery.
3. Patients diagnosed with recurrent ovarian cancer, fallopian cancer, or primary peritoneal cancer who did not receive Bevacizumab chemotherapy
4. Patients with other concurrent disease that can affect overall survival (infection, hypertension, diabetes, cardiac disease, etcetera)
5. Patients with underlying disease (diabetes, neuropathy, brain or bone metastasis) that can induced neuropathy
6. Patients allergic to selenium
7. Inappropriate patients by the researcher's decision

Ages: 19 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2019-12-24 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of chemotherapy-induced peripheral neuropathy (3m) | Examined at 3 months after last paclitaxel chemotherapy
  To evaluate the incidence of CIPN by evaluating paresthesia, pain and motor based on WHO-CIPN criteria.

SECONDARY OUTCOMES:
Incidence of chemotherapy-induced peripheral neuropathy (baseline, 3wk) | Examined on the day 0 of first chemotherapy, 3 weeks after last paclitaxel chemotherapy, and checked before start of every chemotherapy cycles (each cycle is 21 days)
  To evaluate the incidence of CIPN by evaluating paresthesia, pain and motor based on WHO-CIPN criteria.
Severity of chemotherapy-induced peripheral neuropathy | Examined on the day 0 of first chemotherapy, 3 weeks after last paclitaxel chemotherapy, 3 months after last paclitaxel chemotherapy, and checked before start of every chemotherapy cycles (each cycle is 21 days)
  To evaluate the severity of CIPN by evaluating paresthesia, pain and motor based on WHO-CIPN criteria.
Assessment of quality of life1 | Examined on the day 0 of first chemotherapy, 3 weeks after completion of 3 cycles of chemotherapy, 3 weeks after completion of 6 cycles of chemotherapy, and 3 months after completion of 6 cycles of chemotherapy (each cycle is 21 days)
  Scoring of quality of life assessment using European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) Scale: 30-126, the higher score means better quality of life
Assessment of quality of life2 | Examined on the day 0 of first chemotherapy, 3 weeks after completion of 3 cycles of chemotherapy, 3 weeks after completion of 6 cycles of chemotherapy, and 3 months after completion of 6 cycles of chemotherapy (each cycle is 21 days)
  Scoring of quality of life assessment using European Organization for Research and Treatment of Cancer Chemotherapy Induced Peripheral Neuropathy 20 (EORTC-CIPN20) Scale: 20-80, the higher score mean worse symptom
concomitant medication1 | Checked on the day 0 of every cycles of chemotherapy, 3 weeks after completion of 3 cycles of chemotherapy, 3 weeks after completion of 6 cycles of chemotherapy, and 3 months after completion of 6 cycles of chemotherapy (each cycle is 21 days)
  Dosage and usage of concomitant medication (neurontin) for CIPN
concomitant medication2 | Checked on the day 0 of every cycles of chemotherapy (each cycle is 21 days), from day 1 to day 21 on each cycle
  Dosage and usage of concomitant medication (duloxetine) for CIPN
concomitant medication3 | Checked on the day 0 of every cycles of chemotherapy, 3 weeks after completion of 3 cycles of chemotherapy, 3 weeks after completion of 6 cycles of chemotherapy, and 3 months after completion of 6 cycles of chemotherapy (each cycle is 21 days)
  Dosage and usage of concomitant medication (celecoxib) for CIPN
Adverse events 1 | From the day 1 of chemotherapy to the day before starting next cycle (each cycle is 21 days), 3 weeks after completion of 3 cycles of chemotherapy, 3 weeks after completion of 6 cycles of chemotherapy, and 3 months after completion of 6 cycle
  Evaluation of chemotherapy-induced toxicity hematologic (ANC, Hb, Plt) and non-hematologic (nausea, vomiting, diarrhea, constipation, hypersensitivity reaction) symptoms are evaluated by Common Terminology Criteria for Adverse Events ver 5.0 by grade
Adverse events 2 | From the date of first day of chemotherapy to the day before starting next cycle (each cycle is 21 days), 3 weeks after completion of 3 cycles of chemotherapy, 3 weeks after completion of 6 cycles of chemotherapy, and 3 months after completion of 6 cycle
  Evaluation of any toxicity related to intravenous selenium administration (garlic odor, nausea, vomiting, hypersensitivity reaction) symptoms are evaluated by Common Terminology Criteria for Adverse Events ver 5.0 by grade

CONTACTS AND LOCATIONS:
Overall Officials: Hee Seung Kim, MD/PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hay CM, Courtney-Brooks M, Lefkowits C, Hagan TL, Edwards RP, Donovan HS. Symptom management in women with recurrent ovarian cancer: Do patients and clinicians agree on what symptoms are most important? Gynecol Oncol. 2016 Nov;143(2):367-370. doi: 10.1016/j.ygyno.2016.08.235. Epub 2016 Aug 13. PMID 27531571
- [Background] Hausheer FH, Schilsky RL, Bain S, Berghorn EJ, Lieberman F. Diagnosis, management, and evaluation of chemotherapy-induced peripheral neuropathy. Semin Oncol. 2006 Feb;33(1):15-49. doi: 10.1053/j.seminoncol.2005.12.010. PMID 16473643
- [Background] Park SB, Kwok JB, Asher R, Lee CK, Beale P, Selle F, Friedlander M. Clinical and genetic predictors of paclitaxel neurotoxicity based on patient- versus clinician-reported incidence and severity of neurotoxicity in the ICON7 trial. Ann Oncol. 2017 Nov 1;28(11):2733-2740. doi: 10.1093/annonc/mdx491. PMID 29117336
- [Background] Mols F, Beijers T, Vreugdenhil G, van de Poll-Franse L. Chemotherapy-induced peripheral neuropathy and its association with quality of life: a systematic review. Support Care Cancer. 2014 Aug;22(8):2261-9. doi: 10.1007/s00520-014-2255-7. Epub 2014 May 1. PMID 24789421
- [Background] Molassiotis A, Cheng HL, Lopez V, Au JSK, Chan A, Bandla A, Leung KT, Li YC, Wong KH, Suen LKP, Chan CW, Yorke J, Farrell C, Sundar R. Are we mis-estimating chemotherapy-induced peripheral neuropathy? Analysis of assessment methodologies from a prospective, multinational, longitudinal cohort study of patients receiving neurotoxic chemotherapy. BMC Cancer. 2019 Feb 8;19(1):132. doi: 10.1186/s12885-019-5302-4. PMID 30736741
- [Background] Carozzi VA, Canta A, Chiorazzi A. Chemotherapy-induced peripheral neuropathy: What do we know about mechanisms? Neurosci Lett. 2015 Jun 2;596:90-107. doi: 10.1016/j.neulet.2014.10.014. Epub 2014 Oct 22. PMID 25459280
- [Background] Duggett NA, Griffiths LA, McKenna OE, de Santis V, Yongsanguanchai N, Mokori EB, Flatters SJ. Oxidative stress in the development, maintenance and resolution of paclitaxel-induced painful neuropathy. Neuroscience. 2016 Oct 1;333:13-26. doi: 10.1016/j.neuroscience.2016.06.050. Epub 2016 Jul 5. PMID 27393249
- [Background] Erken HA, Koc ER, Yazici H, Yay A, Onder GO, Sarici SF. Selenium partially prevents cisplatin-induced neurotoxicity: a preliminary study. Neurotoxicology. 2014 May;42:71-5. doi: 10.1016/j.neuro.2014.04.002. Epub 2014 Apr 19. PMID 24751598
- [Background] Argyriou AA, Chroni E, Koutras A, Ellul J, Papapetropoulos S, Katsoulas G, Iconomou G, Kalofonos HP. Vitamin E for prophylaxis against chemotherapy-induced neuropathy: a randomized controlled trial. Neurology. 2005 Jan 11;64(1):26-31. doi: 10.1212/01.WNL.0000148609.35718.7D. PMID 15642899
- [Background] Argyriou AA, Chroni E, Koutras A, Iconomou G, Papapetropoulos S, Polychronopoulos P, Kalofonos HP. Preventing paclitaxel-induced peripheral neuropathy: a phase II trial of vitamin E supplementation. J Pain Symptom Manage. 2006 Sep;32(3):237-44. doi: 10.1016/j.jpainsymman.2006.03.013. PMID 16939848
- [Background] Ghoreishi Z, Esfahani A, Djazayeri A, Djalali M, Golestan B, Ayromlou H, Hashemzade S, Asghari Jafarabadi M, Montazeri V, Keshavarz SA, Darabi M. Omega-3 fatty acids are protective against paclitaxel-induced peripheral neuropathy: a randomized double-blind placebo controlled trial. BMC Cancer. 2012 Aug 15;12:355. doi: 10.1186/1471-2407-12-355. PMID 22894640
- [Derived] Yim GW, Han KH, Lee ST, Lee M, Lee SM, Kim HS. Efficacy and safety of intravenous administration of high-dose selenium for preventing chemotherapy-induced peripheral neuropathy in platinum-sensitive recurrent ovarian cancer: a phase 3, double-blind, parallel group, randomized controlled pilot study. BMC Med. 2026 Feb 2. doi: 10.1186/s12916-026-04637-x. Online ahead of print. PMID 41630017
- [Derived] Park SJ, Yim GW, Paik H, Lee N, Lee S, Lee M, Kim HS. Efficacy and safety of intravenous administration of high-dose selenium for preventing chemotherapy-induced peripheral neuropathy in platinum-sensitive recurrent ovarian, fallopian or primary peritoneal cancer: study protocol for a phase III, double-blind, randomized study. J Gynecol Oncol. 2021 Sep;32(5):e73. doi: 10.3802/jgo.2021.32.e73. Epub 2021 Jun 1. PMID 34132071